CLINICAL TRIAL: NCT00243867
Title: A Phase III, Randomized, Study of Weekly Taxoprexin Plus Carboplatin Versus Paclitaxel Plus Carboplatin as First Line Chemotherapy in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Taxoprexin Plus Carboplatin Treatment for Advanced Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-04-20
Record Dates: First submitted 2005-10-21; First posted 2005-10-25 (Estimated); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2018-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — docosahexaenoyl-paclitaxel; Docosahexaenoic Acids; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taxoprexin® and carboplatin (Experimental): Taxoprexin® 400 mg/m² intravenously weekly for 5 weeks
  Carboplatin was given at an Area Under the Curve (AUC) = 4 mg*min/mL on Week 1 and Week 4, Taxoprexin and carboplatin were given up to 3 treatment cycles.
  Interventions: Drug: Taxoprexin; Drug: Carboplatin
- Paclitaxel and carboplatin (Active Comparator): Paclitaxel 225 mg/m² intravenously followed immediately by carboplatin AUC = 6 mg*min/mL. Paclitaxel and carboplatin were given up to 6 treatment cycles.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Taxoprexin — Administered by intravenous infusion over 1 hour infusion
  Other Names: Docosahexaenoic acid (DHA)-paclitaxel
  Arms: Taxoprexin® and carboplatin
Drug: Carboplatin — Administered by intravenous infusion over 30 minutes. Dosing was based on the Calvert formula: carboplatin dose (mg) = (Target AUC) x (glomerular filtration rate (GFR) + 25).
  Other Names: Paraplatin
Drug: Paclitaxel — Administered by intravenous infusion over 3 hour infusion
  Other Names: Taxol
  Arms: Paclitaxel and carboplatin

SUMMARY:
The primary objective of this trial is to compare the survival of patients with advanced non-small cell lung cancer (NSCLC) treated with weekly Taxoprexin in combination with carboplatin to those treated with paclitaxel plus carboplatin in a prospectively randomized trial. In addition, the response rate to each regimen, response duration, time to progression and time to treatment failure will be measured. Toxicity will be evaluated and compared between the two groups.

DETAILED DESCRIPTION:
This is a randomized, multicenter, Phase III open-label study of weekly Taxoprexin® in combination with every three (3) week carboplatin compared to paclitaxel plus carboplatin every three (3) weeks, in patients with advanced non-small cell lung cancer (NSCLC) who have not received cytotoxic agents for advanced disease. Patients may have been previously treated with immunological agents. Patients will be randomized to receive Taxoprexin® at a dose of 400 mg/m2 intravenously by one (1)-hour weekly infusion, 5/6 weeks followed immediately by carboplatin AUC = 4 on weeks one (1) and four (4) as a 30 minute intravenous infusion or paclitaxel 225mg/m2 as a three (3) hour intravenous infusion followed immediately by carboplatin AUC = 6 as a 30 minute intravenous infusion, every three (3) weeks. Patients will receive Taxoprexin® and carboplatin infusions or paclitaxel and carboplatin infusions until progression of disease, intolerable toxicity, completion of six (6) treatment cycles of paclitaxel plus carboplatin or three (3) treatment cycles of Taxoprexin® plus carboplatin, refusal of continued treatment by the patient, or Investigator decision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic or cytologic diagnosis of non-small cell lung cancer. At the time of study entry, patients must have locally advanced (stage IIIb) or metastatic (stage IV) disease.
2. Patients must have at least one site of either measurable or non-measurable disease.
3. Patients must not have received prior systemic chemotherapy for metastatic disease. Prior adjuvant systemic chemotherapy is allowed. At least six (6) months must have elapsed since any prior adjuvant systemic chemotherapy.
4. At least 6 weeks (42 days) since any prior immunotherapy, cytokine, biologic, vaccine or other non chemotherapy anticancer systemic therapies, unless patients have progressed during or after such therapy.
5. At least 4 weeks (28 days) since any prior radiotherapy to > 25% of the bone marrow.
6. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
7. Patients must be at least 18 years of age.
8. Patients must have adequate hepatic and renal function.
9. Patients must have adequate bone marrow function.
10. Life expectancy of at least 3 months.
11. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of their institution.

Exclusion Criteria:

1. Patients who have received prior systemic chemotherapy in the adjuvant setting with a treatment-free interval of less than six (6) months.
2. Patients who have a past or current history of neoplasms other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix and except for other cancers treated for cure and with a disease-free survival greater than 5 years.
3. Patients with symptomatic brain metastasis(es).
4. Women who are pregnant or nursing and men or women who are not practicing an acceptable method of birth control. Women may not breast-feed while on this study.
5. Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
6. Patients with current peripheral neuropathy of any etiology that is greater than grade 1.
7. Patients with unstable or serious concurrent medical conditions.
8. Patients with a known hypersensitivity to Cremophor.
9. Patients with Gilbert's syndrome.
10. Patients must not have had major surgery within the past 14 days.
11. Patients must not receive any concurrent chemotherapy, radiotherapy, or immunotherapy while on study.
12. No known HIV disease or infection.
13. Patients receiving ketoconazole, erythromycin, verapamil, diazepam, quinidine, or diltiazem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falone, MD, Study Director — American Regent, Inc.
Locations (1):
- US Oncology, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Taxoprexin® and Carboplatin: Taxoprexin® 400 mg/m² intravenously weekly for 5 weeks
  Carboplatin was given at an Area Under the Curve (AUC) = 4 mg*min/mL on Week 1 and Week 4, Taxoprexin and carboplatin were given up to 3 treatment cycles.
  Taxoprexin: Administered by intravenous infusion over 1 hour infusion
  Carboplatin: Administered by intravenous infusion over 30 minutes. Dosing was based on the Calvert formula: carboplatin dose (mg) = (Target AUC) x (glomerular filtration rate [GFR] + 25).
- Paclitaxel and Carboplatin: Paclitaxel 225 mg/m² intravenously followed immediately by carboplatin AUC = 6 mg*min/mL. Paclitaxel and carboplatin were given up to 6 treatment cycles.
  Carboplatin: Administered by intravenous infusion over 30 minutes. Dosing was based on the Calvert formula: carboplatin dose (mg) = (Target AUC) x (glomerular filtration rate [GFR] + 25).
  Paclitaxel: Administered by intravenous infusion over 3 hour infusion
Period: Overall Study
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Started | 260 | 258
Completed | 84 | 84
Not Completed | 176 | 174
Not completed — Adverse Event | 24 | 34
Not completed — Lack of Efficacy | 115 | 78
Not completed — Withdrawal by Subject | 11 | 23
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 7
Not completed — Delayed treatment, omission of treatment, peripheral neuropathy, intercurrent illness | 22 | 31

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin | Total
Number analyzed (Participants) | 260 | 258 | 518
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (9.35) | 62.4 (10.54) | 62.8 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 68 | 149
  Male | 179 | 190 | 369
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 249 | 244 | 493
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 161 | 163 | 324
  Russia | 50 | 49 | 99
  Ukraine | 49 | 46 | 95
Disease Stage [Count of Participants; unit: Participants]
  IIIb | 57 | 53 | 110
  IV | 203 | 205 | 408
Weight [Mean (Standard Deviation); unit: kilograms] — Population: One participants weight is missing
  kilograms
    number analyzed (Participants) | 260 | 257 | 517
    (all) | 73.88 (15.111) | 75.46 (17.567) | 74.67 (16.378)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from the day of randomization and ends at death of the participant. Participants were followed every 2 months, whether on or off study, for survival information. Participants alive at the time of termination of the study were considered censored.
Time Frame: Up to 12 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Number analyzed (Participants) | 260 | 258
Months | 8.31 [7.0 to 9.89] | 8.51 [7.82 to 9.69]

2. Secondary Outcome: Percentage of Participants Who Achieved an Objective Complete Response or Partial Response
Description: Antitumor response was defined as the percentage of participants who achieved an objective response (Complete Response or Partial Response), confirmed by repeat assessments performed no less than 4 weeks after the criteria for response were first met. Response was based on the blinded radiological review using Response Evaluation Criteria in Solid Tumors (RECIST) response guidelines, Version 1.0.
  A complete response was defined as a disappearance of all target lesions determined by 2 consecutive observations not less than 4 weeks apart.
  Partial response was defined as a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as reference the baseline sum of LD determined by 2 consecutive observations not less than 4 weeks apart.
Time Frame: Assessed every 6 weeks, up to 12 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Number analyzed (Participants) | 260 | 258
Participants | 40 | 95

3. Secondary Outcome: Duration of Response
Description: Duration of overall response was a measurement from the time measure criteria was met for confirmed complete response or partial response (whichever was first recorded) until the first date that recurrent of progressive disease was objectively documented (taking as reference for progressive disease the smallest measurement recorded since treatment started).
Time Frame: Assessed every 6 weeks, up to 12 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Number analyzed (Participants) | 40 | 95
Months | 5.75 [5.09 to 8.54] | 5.35 [3.98 to 6.21]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the time from randomization to documented disease progression. Progressive disease was defined as at least a 20% increase in the sum of longest diameter (LD) of target lesions, taking as references the smallest sum LD recorded since treatment start or the appearance of 1 or more lesions.
Time Frame: Up to 12 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Number analyzed (Participants) | 260 | 258
Months | 3.02 [2.66 to 4.01] | 4.47 [3.04 to 5.22]

5. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from randomization to the discontinuation of protocol treatment for any reason
Time Frame: Baseline to stopping treatment, up to 12 months
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
Number analyzed (Participants) | 260 | 258
Months | 2.79 [2.10 to 3.02] | 3.25 [2.89 to 3.78]

ADVERSE EVENTS:
Time Frame: Day of initial treatment with study drug until 30 days after last treatment, up to 12 months
Description: An adverse event was defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
  The Safety Set was the population used to evaluate adverse events.
Arm/Group | Taxoprexin® and Carboplatin | Paclitaxel and Carboplatin
All-Cause Mortality (participants affected / at risk) | 198/256 | 196/251
Serious Adverse Events (participants affected / at risk) | 70/256 | 91/251
Other Adverse Events (participants affected / at risk) | 235/256 | 239/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxoprexin® and Carboplatin (N=256) | Paclitaxel and Carboplatin (N=251)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 18 (18)
Dyspenea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
General disorders and administration site conditions (General disorders) | 16 (16) | 19 (19)
Disease progression (General disorders) | 11 (11) | 9 (9)
Asthenia (General disorders) | 2 (2) | 4 (4)
Infections and infestations (Infections and infestations) | 14 (14) | 21 (21)
Infection (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia (Infections and infestations) | 6 (6) | 11 (11)
Cardiac disorders (Cardiac disorders) | 6 (6) | 10 (10)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (7) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (6) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 8 (8)
Nervous system disorders (Nervous system disorders) | 2 (2) | 12 (12)
Vascular disorders (Vascular disorders) | 5 (5) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxoprexin® and Carboplatin (N=256) | Paclitaxel and Carboplatin (N=251)
Fatigue (General disorders) | 101 (101) | 92 (92)
Edema peripheral (General disorders) | 36 (36) | 32 (32)
Asthenia (General disorders) | 29 (29) | 54 (54)
Non-cardiac chest pain (General disorders) | 21 (21) | 23 (23)
Pyrexia (General disorders) | 14 (14) | 13 (13)
Pain (General disorders) | 7 (7) | 14 (14)
Nausea (Gastrointestinal disorders) | 91 (91) | 94 (94)
Constipation (Gastrointestinal disorders) | 63 (63) | 69 (69)
Vomiting (Gastrointestinal disorders) | 37 (37) | 46 (46)
Diarrhea (Gastrointestinal disorders) | 31 (31) | 42 (42)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 18 (18)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 14 (14)
Dyspenia (Respiratory, thoracic and mediastinal disorders) | 56 (56) | 58 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 40 (40)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 6 (6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 11 (11)
Dizziness (Nervous system disorders) | 29 (29) | 29 (29)
Headache (Nervous system disorders) | 25 (25) | 19 (19)
Neuropathy peripheral (Nervous system disorders) | 23 (23) | 54 (54)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (18) | 63 (63)
Dysgeusia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 20 (20)
Neuropathy (Nervous system disorders) | 8 (8) | 23 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (27) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 49 (49)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (18) | 17 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 30 (30)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 13 (13) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 22 (22)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 10 (10)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 17 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (24) | 124 (124)
Rash (Skin and subcutaneous tissue disorders) | 15 (15) | 17 (17)
Anorexia (Metabolism and nutrition disorders) | 38 (38) | 49 (49)
Dehydration (Metabolism and nutrition disorders) | 14 (14) | 29 (29)
Insomnia (Psychiatric disorders) | 28 (28) | 32 (32)
Anxiety (Psychiatric disorders) | 11 (11) | 13 (13)
Depression (Psychiatric disorders) | 9 (9) | 20 (20)
Weight decreased (Investigations) | 19 (19) | 33 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No